CLINICAL TRIAL: NCT01908452
Title: Pyridoxal Kinase Activity in Schizophrenia Patients Without Versus With Tardive Dyskinesia Treated With Vitamin B6
Brief Title: Pyridoxal Kinase Activity in Tardive Dyskinesia
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Not funded
Sponsor: Beersheva Mental Health Center (Other Government)
Collaborators: Sha'ar Menashe Mental Health Center (Other); Tirat Carmel Mental Health Center (Other Government)
Responsible Party: Principal Investigator, Vladimir Lerner, A/Professor, Head of department, Beersheva Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LMRK0911
Record Dates: First submitted 2012-07-25; First posted 2013-07-25 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Tardive Dyskinesia
Keywords: Schizophrenia; pyridoxal kinase activity; plasma pyridoxal level
MeSH Terms: conditions — Tardive Dyskinesia; Schizophrenia | interventions — Pyridoxine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- vitamin B6 (pyridoxine) (Experimental): The 150 participating subjects will be randomized into 2 groups: 75 patients will receive vitamin B6 (1200 mg/day) and 75 patients will receive placebo, each for 12 weeks in a double-blind mode
  Interventions: Drug: Pyridoxine
- placebo (Placebo Comparator): The 150 participating subjects will be randomized into 2 groups: 75 patients will receive vitamin B6 (1200 mg/day) and 75 patients will receive placebo, each for 12 weeks in a double-blind mode
  Interventions: Drug: Pyridoxine

INTERVENTIONS:
Drug: Pyridoxine — 1200 mg/d during 12 weeks

SUMMARY:
Objectives: The mechanisms of tardive dyskinesia (TD) remain unclear, although pathophysiologic theories have proposed mechanisms such as dopamine receptor supersensitivity, the degeneration of cholinergic striatal interneurons, γ-aminobutyric acid (GABA) depletion, and an excess of free radicals.

Prior development of second generation antipsychotic agents, tardive movement disorders were widespread among neuroleptics treated patients. There were great expectations of the new novel drugs. Unfortunately, reports about tardive movement disturbances induced by these medications became more and more frequent, although it has been in use for less than two decades.

A recent study demonstrated that schizophrenic and schizoaffective patients suffering from TD had the mean level of pyridoxal 5'-phosphate (PLP) below lower limit of normal range, while those patients without TD had normal values. At the same time, some open and double-blind placebo-controlled, randomized clinical studies showed that vitamin B6 was very effective in treatment of TD.

Pyridoxal kinase is a key enzyme for the biosynthesis of PLP, the biologically active form of vitamin B6. Some publications reported that the finding of high vitamin B6 levels is consistent with recent reports of low levels of PLP and low activity of pyridoxal kinase. It may explain the functional need for high-dose vitamin B6 supplementation in subjects with TD.

Methods: A multicenter study including 300 schizophrenia and schizoaffective subjects will be performed. The trial will be consisted of 2 parts: the first part a single comparison pyridoxal kinase plasma activity in patients with and without TD; in the second part only TD schizophrenia and schizoaffective patients will continue. It will be a 12-week, randomized, double-blind placebo-controlled trial. Vitamin B6 (1200 mg/day) or placebo capsules will be added to the stable ongoing antipsychotic treatment of 150 schizophrenia patients. Participants will be assessed at baseline and after every 2 weeks of treatment till week 12. Pyridoxal kinase activity will be compared between patients who positively respond to vitamin B6 versus non responders. In addition, PLP levels will be monitored at baseline and at the end of the study.

A battery of research tools will be used for assessment of movement disorders, psychopathology, and side effects. The study will be performed along a period of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients
* DSM-IV diagnosis of schizophrenia or schizoaffective disorder with and without tardive dyskinesia (TD)
* Total ESRS score should be more than 20 in subjects with TD
* Ability to provide a written informed consent

Exclusion Criteria:

* Patients with concurrent medical illness or any movement disorder resemble TD
* Patients who received any vitamin medication
* Evidence of substance or alcohol abuse or a family history of movement disorder.
* Pregnancy and/or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Extrapyramidal Symptom Rating Scale (ESRS) | participants will be followed for the duration of hospital stay every 2 weeks, an expected average of 8 weeks
The Clinical Global Impression Scale (CGI) | participants will be followed for the duration of hospital stay, every 2 weeks. an expected average of 8 weeks
Barnes Akathisia Scale | participants will be followed for the duration of hospital stay, every 2 weeks. an expected average of 8 weeks

SECONDARY OUTCOMES:
The Positive and Negative Syndrome Scale (PANSS) | participants will be followed for the duration of hospital stay, twice during hospitalization. an expected average of 8 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Be'er Sheva Mental Health Center, Beersheba
  - Sha'ar Menashe Mental Health Center, Hadera
  - Tirat Carmel Mental Health Center, Haifa